CLINICAL TRIAL: NCT07312682
Title: Clinical Study on 4DCT-Based Pulmonary Ventilation Imaging for Functional Lung Avoidance in Radiotherapy of Lung Cancer
Brief Title: Application of 4DCT-Based Pulmonary Ventilation Imaging in Lung Cancer Radiotherapy
Acronym: FLAR-4DCT
Status: Active, not recruiting | Type: Observational
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, ZhenZhou Yang, Professor of Radiation Oncology, Cancer Center, Second Affiliated Hospital of Chongqing Medical University, The Second Affiliated Hospital of Chongqing Medical University
Other Study IDs: IRB-2024-394
Record Dates: First submitted 2025-09-09; First posted 2025-12-31 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-12

CONDITIONS: Lung Neoplasms; Radiation Pneumonitis
Keywords: 4DCT; Lung Ventilation Imaging; Functional Lung Imaging; Functional-Lung-Avoidance Radiotherapy (FLAR); IMRT; Organs at Risk (OARs); Radiation-Induced Lung Injury; Radiation Pneumonitis
MeSH Terms: conditions — Lung Neoplasms; Radiation Pneumonitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 4DCT-IMRT Lung Cancer Cohort: Single-center retrospective cohort of consecutive lung cancer patients with high-quality 4DCT planned with IMRT (2022-01-01-2025-09-09; actual enrollment = 202). 4DCT-based ventilation maps delineate high-function lung. Paired-plan comparison of functional-lung-avoidance versus conventional plans; primary outcomes: dose to high-function lung and radiation pneumonitis. Secondary outcomes: doses to heart, spinal cord, and esophagus, and plan-quality metrics (e.g., MLD, V20, DVH). No additional procedures or treatments.

SUMMARY:
This retrospective single-center study investigates whether four-dimensional CT (4DCT)-based lung ventilation imaging can guide functional lung avoidance radiotherapy (FLAR) for patients with primary lung cancer.

Ventilation maps generated from planning 4DCT are used to identify well-ventilated lung regions, enabling paired comparison between functional lung avoidance radiotherapy plans and conventional anatomic radiotherapy plans.

The study aims to assess whether incorporating functional lung information into radiotherapy planning can reduce radiation exposure to well-ventilated lung while maintaining adequate tumor coverage, and to explore its relationship with radiation-induced lung injury.

All analyses are based on existing clinical imaging, treatment planning data, and follow-up records. No additional interventions, imaging, or procedures are performed as part of this study.

DETAILED DESCRIPTION:
This study retrospectively evaluates a functional lung-guided radiotherapy planning workflow based on four-dimensional CT (4DCT) ventilation imaging in patients with primary lung cancer who previously underwent thoracic radiotherapy.

High-quality 4DCT datasets acquired during routine simulation are processed to generate voxel-based lung ventilation maps using deformable image registration and Jacobian-based computational methods. These ventilation maps are spatially registered to planning CT images and incorporated into the treatment planning system to delineate high-function lung subregions.

For each eligible patient, paired radiotherapy plans are retrospectively generated and analyzed: a conventional anatomic radiotherapy plan and a functional lung avoidance radiotherapy (FLAR) plan that incorporates ventilation-defined avoidance structures. Both plans are optimized to achieve comparable target coverage while differing in lung avoidance strategy.

Dosimetric and clinical data are obtained from existing treatment planning records and routine clinical follow-up to support comparative analyses of functional lung sparing and associated pulmonary outcomes. All analyses are conducted retrospectively using data derived from standard clinical care. No prospective enrollment, additional imaging, or study-specific interventions are performed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary lung cancer (adenocarcinoma, squamous cell carcinoma, or small-cell carcinoma) treated with thoracic radiotherapy.
* High-quality 4DCT scans performed before radiotherapy, enabling generation of ventilation or perfusion maps.
* Radiotherapy plans designed using IMRT.
* Availability of both functional lung avoidance plans and conventional anatomical radiotherapy plans for paired analysis.
* Complete treatment and follow-up records, including radiation-induced lung injury (e.g., radiation pneumonitis) and pulmonary function tests.

Exclusion Criteria:

* Incomplete or poor-quality imaging data preventing accurate ventilation/perfusion map generation.
* Radiotherapy interrupted or incomplete for any reason.
* Severe underlying lung diseases (e.g., extensive emphysema, pulmonary fibrosis, active tuberculosis) that may confound treatment outcomes or toxicity assessment.
* Presence of other untreated primary malignancies during the study period.
* Prior lung surgery or local therapies (e.g., ablation) that may affect evaluation of radiation-induced lung injury.
* Missing follow-up data, making assessment of radiation-induced lung injury or long-term lung function changes impossible.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Single-center retrospective cohort of consecutive adults (≥18 years) with primary lung cancer treated with thoracic radiotherapy planned with IMRT, with adequate 4DCT scans for ventilation mapping (2022-01-01 to 2025-09-09).
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2024-12-09 (Actual); Primary Completion 2025-09-09 (Actual); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Radiation-Induced Lung Injury (Grade ≥2) | Assessed at 3 months, 6 months, and 12 months after completion of radiotherapy.
  Incidence of radiation-induced lung injury (RILI) of Grade ≥ 2, assessed using the Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0.
  CTCAE grades range from Grade 1 (mild) to Grade 5 (death related to adverse event), with higher grades indicating more severe toxicity.
  The primary outcome is the proportion of patients experiencing CTCAE Grade ≥ 2 RILI.

SECONDARY OUTCOMES:
Mean Dose to High-Function Lung (Gy) | At baseline treatment planning (prior to radiotherapy delivery).
  DVH-derived mean dose to ventilation-defined high-function lung on paired plans (functional-lung-avoidance vs conventional plans). Lower dose indicates better sparing.
MLD for Whole Lung (Gy) | At treatment planning (baseline, pre-radiotherapy delivery).
  DVH-derived mean lung dose (MLD) for whole lung on paired plans; absolute values reported separately for functional-lung-avoidance vs conventional plans.
V5 of High-Function Lung (%) | At baseline treatment planning (prior to radiotherapy delivery).
  Percentage volume (%) of ventilation-defined high-function lung receiving ≥5 Gy, reported separately for functional-lung-avoidance and conventional radiotherapy plans.
V20 of High-Function Lung | At baseline treatment planning (prior to radiotherapy delivery).
  DVH-derived V20 of ventilation-defined high-function lung, defined as the percentage of lung volume receiving ≥20 Gy, compared between functional-lung-avoidance and conventional radiotherapy plans.
Mean Dose to Heart (Gy) | At treatment planning (baseline, pre-radiotherapy delivery).
  DVH-derived mean dose (Dmean) to the heart, compared between functional-lung-avoidance and conventional radiotherapy plans.
Maximum Dose to Esophagus (Gy) | At treatment planning (baseline, pre-radiotherapy delivery).
  DVH-derived maximum dose (Dmax) to the esophagus, compared between functional-lung-avoidance and conventional radiotherapy plans.
Maximum Dose to Spinal Cord (Gy) | At treatment planning (baseline, pre-radiotherapy delivery).
  DVH-derived maximum dose (Dmax) to the spinal cord, compared between functional-lung-avoidance and conventional radiotherapy plans.
Target Coverage (PTV D95) | At treatment planning (baseline, pre-radiotherapy delivery).
  Percentage of planning target volume (PTV) receiving at least 95% of prescribed dose, compared between functional-lung-avoidance and conventional plans.
Conformity Index of Radiotherapy Plans | At treatment planning (baseline, pre-radiotherapy delivery).
  Conformity Index (CI) of paired treatment plans, comparing functional-lung-avoidance and conventional anatomic radiotherapy plans.
  The Conformity Index is defined as the ratio of the prescription isodose volume to the target volume (CI = V<sub>RI</sub> / V<sub>T</sub>).
  The score ranges from 1.0 to >2.0, where a value closer to 1.0 indicates better conformity and thus higher plan quality.
Homogeneity Index of Radiotherapy Plans | At treatment planning (baseline, pre-radiotherapy delivery).
  Homogeneity Index (HI) of paired treatment plans, comparing functional-lung-avoidance and conventional anatomic radiotherapy plans.
  The Homogeneity Index is defined as (D<sub>2%</sub> - D<sub>98%</sub>) / D<sub>50%</sub>.
  The score typically ranges from 0 to 1.0, where lower values indicate more homogeneous dose distribution and better plan quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center, Second Affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the primary results will be available to qualified researchers upon reasonable request after publication. Available data include demographics, key clinical outcomes (e.g., radiation-induced lung injury), 4DCT-derived ventilation maps, radiotherapy dose/plan files and DVH metrics. Direct identifiers will be removed; data will be shared in compliance with ethics approval and local regulations.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: De-identified IPD and supporting documents will be available from publication of the primary results until 2035-08-31. Requests will be reviewed within 30 days of receipt and, if approved, data will be shared within 60 days after execution of a Data Use Agreement.
Access Criteria: Qualified researchers with a methodologically sound proposal and evidence of IRB/ethics approval may request access. A Data Use Agreement with the sponsor institution is required. Only de-identified data will be shared; no re-identification, redistribution, or commercial use is permitted. Data will be transferred via secure, access-controlled methods. Please contact Zhi Chen (2023440076@stu.cqmu.edu.cn).

REFERENCES:
- [Background] Mattila S, Sovijarvi AR, Harjula A, Viljanen A, Takkunen O, Takkunen H, Mattila I, Mattila P, Merikallio E. Effects of mitral valve replacement on ventilation, volumes, diffusing capacity and regional perfusion of lungs in patients with mitral valve disease. Ann Chir Gynaecol. 1985;74(2):82-5. PMID 3875308
- [Background] Henshaw SK. Induced abortion: a world review, 1990. Fam Plann Perspect. 1990 Mar-Apr;22(2):76-89. PMID 2347411
- [Background] Lombardo J, Castillo E, Castillo R, Miller R, Jones B, Miften M, Kavanagh B, Dicker A, Boyle C, Leiby B, Banks J, Simone NL, Movsas B, Grills I, Guerrero T, Rusthoven CG, Vinogradskiy Y. Prospective Trial of Functional Lung Avoidance Radiation Therapy for Lung Cancer: Quality of Life Report. Int J Radiat Oncol Biol Phys. 2024 Oct 1;120(2):593-602. doi: 10.1016/j.ijrobp.2024.03.046. Epub 2024 Apr 12. PMID 38614278
- See also: National Clinical Research Registration and Filing Information System (China) record for this study(ID：MR-50-25-001899). — https://www.medicalresearch.org.cn/clinicalResearch/researchInfo?id=8d854b86-67c5-4ecb-af5b-ba8120b32339